CLINICAL TRIAL: NCT05278273
Title: A Feasibility Trial and Protocol for Remote Cognitive Training Developed for Use in a Cognitively Healthy Adult Population During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Brian Christie, Professor, University of Victoria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0531
Record Dates: First submitted 2022-03-10; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Cognition Disorders in Old Age
Keywords: 3-dimensional multiple object tracking; Cognitive Training; Neurotracker

STUDY DESIGN:
Intervention Model Description: Twenty adults (10 female, 10 male) will serve as the at-home training group. The cognitive health status for participants will be assessed using a self-report questionnaire and the Mini-Mental State Examination (MMSE), and all participants were deemed cognitively healthy (MMSE > 26). At-home participants loaned the necessary equipment (e.g., 3D-glasses, computer equipment) from the research facilities and engaged in 10 training sessions over five weeks (2x per week). Participant recruitment, retention, adherence and experience will be used as markers of feasibility. For program validation, twenty participants above 50 years old, who had previously completed at least eight sessions of the in-lab 3D-MOT program, were randomly selected as the control group. Individual session scores, overall improvement and learning rates between groups will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At home cognitive training (Experimental): We recruited 20 adults (10 female, mean age = 68.3 years, SD = 6.75) as the at-home training group. We assessed cognitive health status for participants using a self-report questionnaire and the Mini-Mental State Examination (MMSE), and all participants were deemed cognitively healthy (MMSE > 26). At-home participants loaned the necessary equipment (e.g., 3D-glasses, computer equipment) from the research facilities and engaged in 10 training sessions over five weeks (2x per week). Participant recruitment, retention, adherence and experience were used as markers of feasibility.
  Interventions: Device: NeurotrackerX

INTERVENTIONS:
Device: NeurotrackerX — At-home participants loaned the necessary equipment (e.g., 3D-glasses, computer equipment) from the research facilities and engaged in 10 training sessions over five weeks (2x per week). Participant recruitment, retention, adherence and experience were used as markers of feasibility. For program validation, twenty participants above 50 years old, who had previously completed at least eight sessions of the in-lab 3D-MOT program, were randomly selected as the control group.

SUMMARY:
The COVID-19 pandemic has created a shift in the use of at-home spaces for work, play and research. In the current study, the feasibility of implementing an at-home cognitive training tool called NeuroTrackerX, an anaglyph version of the three-dimensional multiple object tracking (3D-MOT) software NeuroTracker was examined, and with the intent of developing an effective protocol and determining the suitability of this tool for research purposes .

DETAILED DESCRIPTION:
The work looks at the feasibility of using a newly developed anaglyph 3D cognitive training tool called NeuroTrackerX in research with adult participants. The work looks to validate an at-home program by comparing participants who complete an online version of Neurotracker (NeurotrackerX) with a group of individuals who completed the classically used in-lab version (Neurotracker). Due to COVID-19, many laboratories forced to transition to remote-based studies, and the purpose of the work is to validate the remote-based protocol. Twenty cognitively healthy adults (10 Male; 10 female) were recruited to engage in this at-home program. The results of these individuals will be compared with results from a group of cognitively healthy adults who had previously engaged in the in-lab version of the program prior to the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for both groups included being aged 50 years and older and to have either normal or corrected vision.

Exclusion Criteria:

* Exclusion criteria included the presence of any major neurocognitive disorder or the presence of visual deficits that impeded one's ability to complete the 3D task.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Neurotracker scores | 5 weeks
  Performance on the multiple-object tracking program across 10 sessions. Scores are between 0 - 4, with increasing scores indicating increasing performance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snowden T, Ohlhauser L, Morrison J, Faubert J, Gawryluk J, Christie BR. A Protocol for Remote Cognitive Training Developed for Use in Clinical Populations During the COVID-19 Pandemic. Neurotrauma Rep. 2023 Aug 14;4(1):522-532. doi: 10.1089/neur.2023.0009. eCollection 2023. PMID 37645472